CLINICAL TRIAL: NCT00242255
Title: Remodeling of Chromatin-Based Epigenetic Structures in Development and Aging
Brief Title: Epigenetics in the Aging Process
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060010; 06-CH-0010
Record Dates: First submitted 2005-10-19; First posted 2005-10-19 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Aging
Keywords: Histone; Chromatin; Epigenome; Senescence; Acetylation; Aging; Tissue Sample

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
This study will examine the role of epigenetics (heritable changes in gene function that occur without a change in DNA sequence) in the aging process. DNA is the primary genetic material, responsible for transmitting information from one cell to the next or from one generation to the next. A second layer of heredity is described by the term "epigenetics."

Epigenetic information is reset from one generation to the next. It works in two ways: 1) by modification of the DNA, like balloons stuck at irregular intervals onto the sides of the DNA helix that encodes genes, and 2) through specialized protein shells that wrap around some regions of DNA. As in DNA, these shells can copy themselves and can transmit instructions. Because they are used to turn genes on and off, errors in their settings cause critical misinformation to be transmitted.

Aging involves many changes, such as muscle weakening, graying hair, skin wrinkling, and so forth. There are several current theories of aging, including damage to genes by oxidation, shortening of tiny structures at the ends of chromosomes called telomeres, and the ability to stretch lifespan with caloric restrictions. This study will investigate the possible role of epigenetics in aging by examining and comparing the shell-like epigenetic settings in skin cells in young adults and older individuals. Preliminary results from earlier studies show differences in these settings in younger and older people.

Women between the ages of 21 and 30 years and 65 and 90 years who are undergoing breast reduction or mastectomy at Suburban Hospital in Bethesda, Maryland, may participate in this study. Tissue removed during surgery for pathological examination will also be used by researchers in this study to validate the preliminary findings noted above and to continue studies into the new area of epigenetics and aging.

...

DETAILED DESCRIPTION:
Normal human lifespan is marked by a complex series of developmental events, relative stability during adulthood, and ultimately a gradual decline in viability. Biological clocks presumably underlie the developmental events that occur through childhood and adolescence, but the nature of those clocks has remained obscure. Progress in this area would be of considerable importance, not only for our understanding of child development, but also because instability in putative clock-like mechanisms may occur as part of the aging process. Such instability could well compromise tissue function and contribute to many of the common degenerative diseases of later life. We propose to investigate whether developmental clocks and related aspects of the aging process are attributable in part to age-related epigenome remodeling. Experiments done to date with cultured human fibroblasts derived from tissue banks provide tentative support for this hypothesis. To exclude tissue culture-related artifacts and to continue the work, it is essential to have access to fresh tissue material in the form of surgically obtained skin specimens that would otherwise be discarded. Elective breast reduction mammoplasty is a frequently performed surgery at Suburban Hospital, Bethesda, Maryland. Small skin specimens will be obtained from this procedure, as well as from normal skin derived from mastectomies. Patients who are to undergo these procedures will be asked to sign a consent form allowing the specimens, normally discarded, to be used instead for research on the mechanism of aging. They will be informed that clinical information will accompany the specimens, including age and known disease conditions. Twenty patients in each of two age ranges, 21-30 yr and 65-90 yr, will be enrolled in the study. The primary outcome will be confirmation of age-related epigenome change in the chromosome 4q35.2 region, previously documented using tissue bank-derived cultured skin fibroblasts. Mapping and sampling chromatin from this region revealed higher histone H4 acetylation in young (24-30 yr) than old (80-85 yr) individuals. Confirmation of this change in primary fibroblasts will be followed by more detailed mapping of chromatin structure and extension beyond the currently defined limits. Secondary outcomes will include examination of two areas of epigenome remodeling that appear to occur between birth and adulthood, as well as searches for additional regions of age-related chromatin change.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 21-30 or 65-90, female or male

Normal liver function, renal function adjusted for age

Written informed consent

EXCLUSION CRITERIA:

Down's or other premature aging syndromes

Mastectomies: skin involvement in the malignant process or damage due to prior radiation therapy

Active skin infection

Skin damage due to photoaging will be noted but will not be a basis for exclusion

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Neonatal cord blood samples collected in association with normal deliveries at a NICHD obstetrics service in Wayne State University (PI Dr. Roberto Romero). Adult samples collected from volunteers at the NIH Blood Bank.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-09-23 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Improved understanding of dynamic epigenome change and its roles in development and aging | Cross-sectional study design with measures corresponding to collection time point
  Publication of scholarly articles describing previously unknown modes of postnatal human epigenome change and their consequences for gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H Howard, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (4):
- United States (4):
  - GW University Medical Center, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Balaban RS, Nemoto S, Finkel T. Mitochondria, oxidants, and aging. Cell. 2005 Feb 25;120(4):483-95. doi: 10.1016/j.cell.2005.02.001. PMID 15734681
- [Background] Bandyopadhyay D, Medrano EE. The emerging role of epigenetics in cellular and organismal aging. Exp Gerontol. 2003 Nov-Dec;38(11-12):1299-307. doi: 10.1016/j.exger.2003.09.009. PMID 14698809
- [Background] Bestor TH. The DNA methyltransferases of mammals. Hum Mol Genet. 2000 Oct;9(16):2395-402. doi: 10.1093/hmg/9.16.2395. PMID 11005794
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-CH-0010.html